CLINICAL TRIAL: NCT04758273
Title: Evaluation of the Safety and Immunogenicity of Inactivated SARS-CoV-2 Vaccine (Vero Cells) in Healthy Population Aged 18 Years and Above: a Randomized, Double-blind, Placebo Parallel-controlled Phase I Clinical Trial
Brief Title: A Safety and Immunogenicity Study of Inactivated SARS-CoV-2 Vaccine (Vero Cells) in Healthy Population Aged 18 Years and Above(COVID-19)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Collaborators: Shenzhen Kangtai Biological Products Co., LTD (Industry); Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020L001-1A
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- medium dosage on day 0, 14(18~59 years) (Experimental): Two doses of medium dosage inactivated SARS-CoV-2 vaccine on the schedule of day 0,14
  Interventions: Biological: medium dosage inactivated SARS-CoV-2 vaccine
- high dosage on day 0, 14(18~59 years) (Experimental): Two doses of high dosage inactivated SARS-CoV-2 vaccine on the schedule of day 0,14
  Interventions: Biological: high dosage inactivated SARS-CoV-2 vaccine
- placebo on day 0, 14(18~59years) (Placebo Comparator): Two doses of placebo on the schedule of day 0,14
  Interventions: Biological: Placebo
- medium dosage on day 0, 28, 56(18~59 years) (Experimental): Three doses of medium dosage inactivated SARS-CoV-2 vaccine on the schedule of day 0,28,56
  Interventions: Biological: medium dosage inactivated SARS-CoV-2 vaccine
- high dosage on day 0, 28, 56(18~59 years) (Experimental): Three doses of high dosage inactivated SARS-CoV-2 vaccine on the schedule of day 0,28,56
  Interventions: Biological: high dosage inactivated SARS-CoV-2 vaccine
- placebo on day 0, 28, 56(18~59 years) (Placebo Comparator): Three doses of placebo on the schedule of day 0,28,56
  Interventions: Biological: Placebo
- medium dosage on day 0, 28, 56(>59 years) (Experimental): Three doses of medium dosage inactivated SARS-CoV-2 vaccine on the schedule of day 0,28,56
  Interventions: Biological: medium dosage inactivated SARS-CoV-2 vaccine
- high dosage on day 0, 28, 56(>59 years) (Experimental): Three doses of high dosage inactivated SARS-CoV-2 vaccine on the schedule of day 0,28,56
  Interventions: Biological: high dosage inactivated SARS-CoV-2 vaccine
- placebo on day 0, 28, 56(>59 years) (Placebo Comparator): Three doses of placebo on the schedule of day 0,28,56
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: medium dosage inactivated SARS-CoV-2 vaccine — medium dosage
  Arms: medium dosage on day 0, 14(18~59 years); medium dosage on day 0, 28, 56(18~59 years); medium dosage on day 0, 28, 56(>59 years)
Biological: high dosage inactivated SARS-CoV-2 vaccine — high dosage
  Arms: high dosage on day 0, 14(18~59 years); high dosage on day 0, 28, 56(18~59 years); high dosage on day 0, 28, 56(>59 years)
Biological: Placebo — placebo
  Arms: placebo on day 0, 14(18~59years); placebo on day 0, 28, 56(18~59 years); placebo on day 0, 28, 56(>59 years)

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase Ⅰ clinical trial of the SARS-CoV-2 inactivated vaccine to evaluate the safety and immunogenicity of the experimental vaccine in healthy adults ⩾18 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy permanent residents aged 18 years and above;
2. Subjects agree to sign the informed consent forms voluntarily;
3. Subjects are able to comply with the requirements of the clinical trial protocol;
4. Armpit temperature <=37.0 degree C;
5. Female subjects of childbearing age were not pregnant at the time of enrollment, were not breastfeeding, and had no birth plan within the first 3 months after enrollment; effective contraceptive measures had been taken within 2 weeks before enrollment.

Exclusion Criteria:

1. Within 14 days before vaccination, subjects have been abroad and to villages/communities experienced COVID-19 epidemics, and in contact with COVID-19 cases or suspected cases. Subjects are under isolation observation, or living in the villages/communities with COVID-19 cases or suspected cases;
2. Confirmed cases, suspected cases or asymptomatic cases with COVID-19 (refer to Information System of China Disease Prevention and Control);
3. Subjects with history of SARS virus infection by self-reported;
4. Positive in throat swab through RT-PCR;
5. Positive in SARS-CoV-2 antibody test;
6. Subjects with abnormal indicators, such as blood biochemistry, blood routine, urine routine and coagulation function which might show clinical meaning, before administration;
7. Subjects with history of severe allergic reactions (such as acute anaphylaxis, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain) or allergy to known composition of inactivated SARS-CoV-2 vaccine;
8. Subjects with history of convulsion, epilepsy, encephalopathy or mental illness or family history;
9. Subjects with congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
10. Subjects with known or suspected diseases include: severe respiratory diseases, severe cardiovascular diseases, severe liver and kidney diseases, uncontrollable hypertension (systolic pressure >=140 mmHg, diastolic pressure >=90 mmHg; subjects aged >=60 years with systolic pressure >=150 mmHg, diastolic pressure >=100 mmHg), diabetic complications, malignant tumors, various acute diseases or acute onset of chronic diseases;
11. Subjects diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
12. Subjects with history of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease);
13. Subjects receiving anti-TB treatment;
14. Subjects receiving other research drugs within 6 months before vaccination;
15. Subjects receiving immunotherapy or inhibitor therapy within 3 months (consistently oral or infusion for more than 14 days);
16. Subjects receiving blood products within 3 months before administration;
17. Subjects vaccinated with live attenuated vaccine within 14 days before vaccination;
18. Subjects vaccinated with other vaccine within 7 days before vaccination;
19. The researchers shall judge the other conditions which might be not in compliance with the requirements of this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions/events | 0-28 days after each dose of vaccination

SECONDARY OUTCOMES:
Serious Adverse Events (SAE) | within 12 months post full vaccination
Incidence of abnormal indicators of laboratory safety examinations(including blood routine, blood biochemistry, urine routine and coagulation function) | Day 3 after each dose of vaccination
The seropositive rates of SARS-CoV-2 neutralizing antibody | Day 14 and day 28 after each dose of vaccination, and 3, 6 and 12 months post full vaccination
The seropositive level of SARS-CoV-2 neutralizing antibody | Day 14 and day 28 after each dose of vaccination, and 3, 6 and 12 months post full vaccination
The seropositive rates of SARS-CoV-2 IgG antibody(tested by ELISA) | Day 14 and day 28 after each dose of vaccination, and 3, 6 and 12 months post full vaccination
The seropositive level of SARS-CoV-2 IgG antibody(tested by ELISA) | Day 14 and day 28 after each dose of vaccination, and 3, 6 and 12 months post full vaccination
The proportion of IFN-γ positive cells (by ELISpot) | Before second and third vaccination, day 28 post full vaccination(18~59years, 3 doses group); before second vaccination and day 14 post full vaccination(18~59years, 2 doses group); 3, 6 and 12 months post full vaccination(18~59years, both group）
Level of IL-2、IL-4、IL-5、IL-6、TNFα、IFN-γ (by ELISA) | Before second and third vaccination, day 28 post full vaccination(18~59years, 3 doses group); before second vaccination and day 14 post full vaccination(18~59years, 2 doses group); 3, 6 and 12 months post full vaccination(18~59years, both group）

OTHER OUTCOMES:
The SARS-CoV-2 antibody level of IgG1, IgG2, IgG3, IgG4 and Nucleoprotein | Day 14 and 28 after each dose, and 3, 6, 12 months post full vaccination(18~59years)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China